CLINICAL TRIAL: NCT01288261
Title: A Phase I Trial of Weekly Paclitaxel in Combination With Bavituximab in Patients With Her-2 Negative Metastatic Breast Cancer
Brief Title: Paclitaxel and Bavituximab in Treating Patients With HER2-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0884-04; NCI-2011-00026 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA023074 (NIH)
Record Dates: First submitted 2011-01-27; First posted 2011-02-02 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Male Breast Cancer; Recurrent Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Paclitaxel; Taxes; bavituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Paclitaxel, bavituximab, laboratory biomarker analysis and pharmacological study
  Interventions: Drug: paclitaxel; Biological: bavituximab; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: bavituximab — Given IV
  Other Names: Tarvacin
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative study
  Other Names: pharmacological studies

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bavituximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving paclitaxel together with bavituximab may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of giving paclitaxel and bavituximab together in treating patients with Human Epidermal growth factor Receptor 2 (HER2 )-negative metastatic breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, feasibility, and tolerability of combining paclitaxel with weekly bavituximab therapy.

SECONDARY OBJECTIVES:

I. To describe changes in pharmacodynamic markers and coagulation markers in response to single agent and combined therapy.

OUTLINE:

Patients receive paclitaxel intravenously (IV) on days 1, 8, and 15 and bavituximab IV on days 1, 8, 15, and 22 (days 15 and 22 only of course 1). Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained
* Life expectancy of at least 3 months
* Histologically or cytologically confirmed, Her-2 negative breast cancer with evidence of metastatic disease
* Measurable or evaluable disease by Response Evaluation Criteria In Solid Tumors (RECIST)
* Eastern Cooperative Oncology Group (ECOG) Performance Status =< 2
* Adequate hematologic function (absolute neutrophil count [ANC] >= 1,500 cells/uL; hemoglobin >= 9 g/dL; platelets >= 100,000/uL and =< 500,000/uL)
* Adequate renal function (serum creatinine =< 1.5 mg/dL or calculated creatinine clearance >= 60 ml/min)
* Adequate hepatic function (total or direct bilirubin =< Upper Limit of Normal (ULN), Alk Phos =< 4 x ULN)
* Prothrombin time international normalized ratio within institutional normal limits
* Activated partial thromboplastin time =< 1.5 x ULN
* New York Heart Association classification I or II
* Female patients must have a negative urine pregnancy test at prestudy (not applicable to patients with bilateral oophorectomy and/or hysterectomy or to those patients who are postmenopausal)

Exclusion Criteria:

* Known history of bleeding diathesis or coagulopathy (e.g., von Willebrand Disease, Hemophilia)
* Any current evidence of clinically significant active bleeding
* Any history of significant thromboembolic events (i.e., deep vein thrombosis or pulmonary thromboembolism) within the last five years or requirement for ongoing therapy with oral or parenteral anticoagulants; central venous catheter-related thrombosis > 12 months ago and low dose anticoagulants to maintain patency of lines are allowed; patients taking anticoagulants (e.g., prophylactic heparin or enoxaparin) are required to observe the washout period of 1 week prior to study drug infusion on Study Day 1
* Concurrent hormone therapy (i.e., estrogen contraceptives, hormone replacement, anti-estrogen); patients taking concurrent hormone therapy are required to observe the washout period of 2 weeks prior to study drug infusion on Study Day 1
* Grade 2 or higher peripheral neuropathy (e.g., numbness, tingling, and/or pain in distal extremities)
* More than one prior chemotherapy regimen for metastatic disease (prior adjuvant chemotherapy or any number of prior hormonal therapies are allowed)
* Chemotherapy, immunotherapy or radiotherapy within 2 weeks of Study Day 1 or not having recovered from significant treatment-related side effects due to agents administered previously; patients who have receive nitrosoureas and mitomycin C therapy are required to observe the washout period of 6 weeks prior to study drug infusion on Study Day 1
* Allergy to polysorbate 80 or drugs containing polyoxyethylated castor oil (e.g. cyclosporine)
* Symptomatic or clinically active Central Nervous System (CNS) disease
* Major surgery within 4 weeks of Study Day 1
* Female patients pregnant or nursing
* All patients of reproductive potential must agree to use appropriate non-hormonal form of contraception
* Uncontrolled intercurrent disease (e.g., diabetes, hypertension, thyroid disease)
* Any history of angina pectoris, coronary artery disease or cerebrovascular accident, or transient ischemic attack
* A history of any condition requiring anti-platelet therapy (e.g., phosphodiesterase inhibitors, adenosine diphosphate receptor antagonists) with the exception of general cardiovascular prophylaxis with aspirin
* Cardiac arrhythmia requiring medical therapy
* Serious non-healing wound (including wound healing by secondary intention, ulcer, or bone fracture)
* Requirement for chronic daily steroid use
* Known chronic infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Determination of grade 3 or higher toxicities associated with the combination therapy as classified using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | One year

SECONDARY OUTCOMES:
Overall response rate of the regimen by RECIST | One year
Progression free survival (PFS) | One year
Measurable changes in levels of circulating endothelial cells (CEC), circulating endothelial progenitors (CEP), apoptotic CEC, and circulating tumor cells (CTC), as well as changes in cell-specific microparticle formation in response to therapy | One year
Activation of coagulation as measured by changes in D-dimer levels and platelet activation markers in response to therapy | One year
Collection and storage of additional plasma for further analysis of angiogenic markers (i.e., VCAM and VEGF) | One year

CONTACTS AND LOCATIONS:
Overall Officials: Alison Stopeck, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States